CLINICAL TRIAL: NCT06591130
Title: A Pilot Trial of a Culturally Adapted Intervention to Prevent Self-harm in Young People With Autism
Brief Title: Culturally Adapted Intervention to Prevent Self-harm in Young People With Autism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OAR-ASD-002
Record Dates: First submitted 2024-08-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder; Self Harm
Keywords: Autism; Self harm; Youth suicidality
MeSH Terms: conditions — Autism Spectrum Disorder; Self-Injurious Behavior; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-CMAP + TAU (Experimental)
  Interventions: Behavioral: Youth culturally adapted manual assisted psychological intervention (Y-CMAP)
- TAU alone (No Intervention): Treatment as usual (TAU) will include standard routine care that participants could potentially be receiving by their treating GP, or from autism centers, such as behavioral therapy, psychoeducation, occupational therapy, sports therapy, and art therapy. We will maintain a detailed record of each participant's routine care.

INTERVENTIONS:
Behavioral: Youth culturally adapted manual assisted psychological intervention (Y-CMAP) — YCMAP (Youth culturally adapted manual assisted psychological intervention) is based on CBT principles. It comprises of 8-10 sessions delivered individually over 3 months (weekly for 1 month then fortnightly), lasting for 60 minutes. The intervention includes psycho-education and a comprehensive cognitive behavioural assessment of the self-harm attempt using virtual stories of four young people. Therapists and young person choose from a list of techniques those which are most relevant to the young person's problems. Therapy is therefore adapted to fit with the young person's problems and primarily utilises problem solving, CBT, and dialectical therapy strategies to bring about change. To help determine the most appropriate coping strategy a coping tree is designed. Training in assertiveness and anger management are offered to help the young person to develop resilience to cope with stress.
  Arms: Y-CMAP + TAU

SUMMARY:
The goal of this feasibility randomized controlled trial is to assess the feasibility and acceptability of Youth Culturally Adapted Manually Assisted brief psychological intervention (YCMAP) in young people with autism in Pakistan. In a rater-blind, 2-arm, multi-site, feasibility randomized controlled trial (RCT), participants will be randomized either to 1) YCMAP added to the Treatment as Usual (TAU) or 2) TAU alone. Participants in the Y-CMAP arm will receive 8-10 sessions delivered individually over 3 months (weekly for 1 month then fortnightly), lasting for 60 minutes. Assessments will be conducted at baseline and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-24 years
* History of self-harm and/or possible suicidal behavior
* Able to engage in assessment and intervention
* Ability to provide informed consent

Exclusion Criteria:

* Young people with autism with limited receptive and expressive language skills that would prevent engagement
* With any chronic medical disorder or physical condition (including communicable diseases such as Tuberculosis) that would prevent participation in assessments and or intervention.
* Not willing to participate.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility | Baseline to 12 weeks
  Data on recruitment and retention rates. The success criterion of feasibility will be to recruit > 50% of eligible participants and retain 70%.
Intervention acceptability | Baseline to 12 weeks
  Acceptability will be assessed using data on attendance. The criterion for acceptability is the mean attendance rate of >70% of sessions.

SECONDARY OUTCOMES:
Suicide Attempt and Self-Harm | Baseline to 12 weeks
  This consists of four questions measuring the previous suicide attempt and the presence of self-harm. The scale was taken from the original Self-Harm Questionnaire.
Beck Scale for Suicide Ideation | Baseline to 12 weeks
  A 19-item instrument for detecting and measuring the current intensity of patient-specific attitude, behavior, and specificity of patient thoughts to kill him/ herself during the past week.
Card sort Task for Self-harm Behavior | Baseline to 12 weeks
  117 cards related to thoughts, feelings, events, behaviours and self-harm supports/services
Beck Hopelessness Scale | Baseline to 12 weeks
  This instrument is designed to measure three aspects of hopelessness, feelings about the future, loss of motivation and expectations.
Autistic Depression Assessment Tool - Adult | Baseline to 12 weeks
  It has 21 items capturing depression symptoms in the past 14 days. The Autistic Depression Assessment Tool - Adult has staged questions for each symptom: 1) the presence (yes/no) of the difficulty in the past 14 days; 2) if present, the length of time the difficulty has been experienced for over the past 14 days (from 1-3 days (1) to 12-14 days (4)); and 3) the impact of the symptom on everyday functioning (from "Never" (0) to "Extremely" (4)). Answering "no" to a difficulty is scored 0, length of time is scored from 1-4, and impact from 1-4. Scores across the sections are summed to obtain individual item scores from 0-8, with total scores ranging from 0-168, with higher scores indicating a greater number / impact of depressive symptoms in the past 14 days.
Kessler Psychological Distress Scale | Baseline to 12 weeks
  The Kessler Psychological Distress Scale is a simple measure of psychological distress. The scale involves 10 questions about emotional states each with a five-level response scale. The measure can be used as a brief screen to identify levels of distress. Each item is scored from one 'none of the time' to five 'all of the time'. Scores of the 10 items are then summed, yielding a minimum score of 10 and a maximum score of 50. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress.
Euro-Qol-5 Dimensions scale | Baseline to 12 weeks
  It's a standardised instrument to measure participants' health-related quality of life. It consists of a self-report questionnaire covering five dimensions of health (mobility, self-care, usual activities, pain/ discomfort, and anxiety/ depression)
Autism Diagnostic Observation Schedule | Baseline
  Autism Diagnostic Observation Schedule is a semi-structured, standardized assessment measuring social interaction, communication, play, and imaginative use of materials for individuals suspected of experiencing ASD. It consists of four different modules as per the age and expressive language, from preverbal children to verbally proficient adults. Behaviours are coded in the areas of social communication, social relatedness, play and imagination, and restricted interests and repetitive behaviours. Internal consistency ranges from 0.47 to 0.94 for all domains and modules ranges from 0.47 to 0.94.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, FRCPsych, Principal Investigator — Pakistan Institute of Living and Learning

IPD SHARING:
Plan to Share IPD: No